CLINICAL TRIAL: NCT05805670
Title: Feasibility of Implementing Yoga and Meditation in the Preoperative Period of Pediatric Idiopathic Scoliosis Surgery, an Exploratory Study
Brief Title: Preoperative Yoga and Meditation for Pediatric Idiopathic Scoliosis Surgery
Acronym: YOMEPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0057
Record Dates: First submitted 2023-02-27; First posted 2023-04-10 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Juvenile and Adolescent Idiopathic Scoliosis
Keywords: Yoga; Meditation; Mindfulness; Anesthesia; Idiopathic Scoliosis Surgery; Anxiety; Children; Pediatric
MeSH Terms: conditions — Anxiety Disorders | interventions — Yoga; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with surgical indication scoliosis follow the Yoga and Mindfulness protocol before surgery (Experimental): Intervention is a noninvasive approach. The protocol is composed of 5 sessions containing simple yoga postures and meditation audio supports to listen to.
  Interventions: Other: Yoga and Mindfulness

INTERVENTIONS:
Other: Yoga and Mindfulness — Intervention is a noninvasive approach. The protocol is composed of 5 sessions containing simple yoga postures and meditation audio supports to listen to and 1 post-operative visit (24 hours after surgery)
  The 5 sessions will be carried out 1 session/week from inclusion to the day before surgery

SUMMARY:
This study has to purpose Yoga and Meditation before surgery for idiopathic scoliosis.

Protocol's observance will tell the investigators if it is feasible and appropriate in a University hospital center.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis is the most common deforming orthopedic condition.

Preoperative anxiety is increased by operating time, post-operative pain level, neurological and hemorrhagic risk.

The aim of the study was to purpose five sessions of Yoga and Meditation before surgery, remotely and face-to-face.

Observance of the 5 sessions will tell us if this protocol is feasible and appropriate. Preoperative anxiety intensity will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age from 8 to 17 years
* Female and male gender
* Planned idiopathic scoliosis surgery

Exclusion Criteria:

* Physical inability to do simple yoga postures during the initial session
* Neurological spinal deformity (cerebral palsy, severe epileptic disease, myopathy)
* Misunderstanding of the french language
* Recent history of characterized depressive episode: hospitalization and/or antidepressant treatment in the last 6 months
* Time between the first YOMEPOP session and the date of the operation less than 28 days
* Refusal of permission to take picture
* Failure to obtain informed consent from one of the parents with parental authority
* Absence of affiliation to a French social security scheme or beneficiary of such a scheme
* Patient with a legal protection measure

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-03-16 (Actual); Study Completion 2024-03-16 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with observance greater than or equal to 2 | During the preoperative period
  Yoga and Meditation protocol's observance will be rated from 0 to 3 (0 is a session not completed to 3 is a fully completed session)

SECONDARY OUTCOMES:
VAS-anxiety scores | From preoperative period up to 1 day postoperative
  To evaluate the level of anxiety thanks to Visual Analogue Scale (VAS) The VAS-anxiety is rated from 0 to 10
FPS-R scores | From preoperative period up to 1 day postoperative
  To evaluate the level of pain thanks to Face Pain Scale-Revised (FPS-R) The FPS-R scale is rated from 0 to 10 (0 is no pain to 10 extreme pain)
Assessment of satisfaction of Yoga and Meditation protocol | The day before the surgery
  Satisfaction of parents and child will be rated from 1 to 3
  1. Not satisfied
  2. Moderately satisfied
  3. Satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle VEISLINGER, Principal Investigator — Hospital of Montpellier
Locations (1):
- UH of Montpellier, Montpellier, France